CLINICAL TRIAL: NCT04016272
Title: Self-Administered Transcranial Direct Current Stimulation for Pain in Older Adults With Knee Osteoarthritis: A Phase II Randomized Sham-Controlled Trial
Brief Title: Self-Administered Transcranial Direct Current Stimulation for Pain in Older Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hyochol Ahn, PhD, Associate Dean for Research & Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-SN-19-0469; R15NR018050 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: Active tDCS
- Sham tDCS (Placebo Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — tDCS with a constant current intensity of 2 mA will be applied for 20 minutes per session daily for 2 weeks (Monday to Friday) via the Soterix 1x1 tDCS mini-CT Stimulator device (Soterix Medical Inc., NY) with headgear and saline-soaked surface sponge electrodes.
  Other Names: Soterix 1x1 tDCS mini-CT Stimulator
  Arms: Active tDCS
Device: Sham tDCS — For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds.
  Other Names: Soterix 1x1 tDCS mini-CT Stimulator
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and efficacy of self-administered transcranial direct current stimulation (tDCS) in older adults with knee osteoarthritis (OA)

ELIGIBILITY:
Inclusion Criteria:

* have symptomatic knee OA based on American College of Rheumatology Clinical criteria
* have had knee OA pain in the past 3 months with an average of at least 30 on a 0-100 NRS for pain
* can speak and read English
* have no plan to change medication regimens for pain throughout the trial

Exclusion Criteria:

* prosthetic knee replacement or nonarthroscopic surgery to the affected knee
* history of brain surgery, brain tumor, seizure, stroke or intracranial metal implantation
* systemic rheumatic disorders, including rheumatoid arthritis, systemic lupus erythematosus, and fibromyalgia
* alcohol/substance abuse
* current use of sodium channel blockers, calcium channel blockers and NMDS receptor antagonists
* diminished cognitive function that would interfere with understanding study procedures(i.e., Mini-Mental Status Exam score ≤ 23)
* pregnancy or lactation
* hospitalization within the preceding year for psychiatric illness
* no access to a device with internet access that can be used for secure videoconferencing for real-time remote supervision

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, PhD, RN, MSN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee C, Park J, Kwoh CK, Fain M, Park L, Ahn H. Home-Based, Remotely Supervised Transcranial Direct Current Stimulation Improves the Overall Pain Experience of Older Adults With Knee Osteoarthritis. Pain Res Manag. 2025 Feb 24;2025:1783171. doi: 10.1155/prm/1783171. eCollection 2025. PMID 40040747
- [Derived] Park J, Tong H, Kang Y, Miao H, Lin L, Fox RS, Telkes I, Martorella G, Ahn H. Comparison of responders and nonresponders with knee osteoarthritis after transcranial direct current stimulation. Pain Manag. 2024 Sep;14(9):507-518. doi: 10.1080/17581869.2024.2429943. Epub 2024 Nov 16. PMID 39548963
- [Derived] Martorella G, Mathis K, Miao H, Wang D, Park L, Ahn H. Self-administered transcranial direct current stimulation for pain in older adults with knee osteoarthritis: A randomized controlled study. Brain Stimul. 2022 Jul-Aug;15(4):902-909. doi: 10.1016/j.brs.2022.06.003. Epub 2022 Jun 8. PMID 35690388

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS: tDCS with a constant current intensity of 2 mA was applied for 20 minutes five times a week (Monday to Friday) for 3 weeks via the Soterix 1 × 1 tDCS mini-CT Stimulator device (Soterix Medical Inc., New York, NY, USA; 6.5 inches long, 3 inches wide, 0.7 inches thick) with headgear and 5 × 7 cm sponge electrodes.
- Sham tDCS: tDCS with a constant current intensity of 2 mA was applied for 30 seconds out of 20 minutes five times a week (Monday to Friday) for 3 weeks via the Soterix 1 × 1 tDCS mini-CT Stimulator device (Soterix Medical Inc., New York, NY, USA; 6.5 inches long, 3 inches wide, 0.7 inches thick) with headgear and 5 × 7 cm sponge electrodes.
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 61 | 62
Completed | 60 | 60
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: We analyzed the data from subjects who completed the study only.
Groups:
- Active tDCS: 2mA current is applied for 20 minutes.
- Sham tDCS: 2mA current is applied for 30 seconds.
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.32 (8.41) | 66.60 (8.43) | 65.96 (8.407)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 53 | 56 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 22 | 41
  White | 33 | 36 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Pain as Assessed by the Numeric Rating Scale (NRS) for Pain
Description: The Numeric Rating Scale (NRS) total score ranges from 0 (no pain) to 100 (most intense pain imaginable).
Time Frame: baseline, week 3
Population: Comparison of pain intensity changes between two groups at 3 weeks from baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 60 | 60
score on a scale | -24.07 (21.55) | -1.08 (16.46)

2. Secondary Outcome: Change in Pain Related Cortical Response Using a Continuous Wave, Multichannel Functional Near-infrared Spectroscopy (fNIRS) Imaging System
Description: Pain-related cortical response will be measured using a continuous-wave, multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) with three semiconductor lasers at 780, 805, and 830 nm. Optical recordings will be collected during thermal and punctate pain stimulation and correlation values will be presented in the form of figures.
  * Specify the full scale: Pearson correlation coefficient (r) between pairs of brain regions (fNIRS channels).
  * A value of r=0 indicates that two brain regions were functionally disconnected.
  * Greater absolute r values denote stronger connections. However, this does not indicate a better or worse result but only a different type of connectivity on a macroscale (when considering several fNIRS channels).
  * We used |r|>0.3 (absolute value of r greater than 0.3) to extract meaningful functional connections.
Time Frame: Baseline, week1, week2, and week 3
Population: All Subjects completed fNIRS.
Measure: Mean (Standard Deviation); unit: Pearson correlation coefficient
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 61 | 62
Pearson correlation coefficient
  Connectivity within Primary motor-somatosensory cortices at baseline | 0.18 (0.21) | 0.12 (0.17)
  Connectivity within Prefrontal cortex at baseline | 0.10 (0.12) | 0.09 (0.11)
  Connectivity between PFC and M1_S1 cortices at baseline | -0.12 (0.17) | -0.12 (0.16)
  Connectivity within Primary motor-somatosensory cortices at week 1 | 0.17 (0.20) | 0.14 (0.18)
  Connectivity within Prefrontal cortex at week 1 | 0.09 (0.13) | 0.16 (0.15)
  Connectivity between PFC and M1_S1 cortices at week 1 | -0.13 (0.12) | -0.17 (0.17)
  Connectivity within Primary motor-somatosensory cortices at week 2 | 0.17 (0.17) | 0.14 (0.19)
  Connectivity within Prefrontal cortex at week 2 | 0.09 (0.09) | 0.10 (0.11)
  Connectivity between PFC and M1_S1 cortices at week 2 | -0.14 (0.13) | -0.15 (0.20)
  Connectivity within Primary motor-somatosensory cortices at week 3 | 0.18 (0.14) | 0.17 (0.14)
  Connectivity within Prefrontal cortex at week 3 | 0.10 (0.11) | 0.10 (0.10)
  Connectivity between PFC and M1_S1 cortices at week 3 | -0.14 (0.10) | -0.17 (0.15)

3. Secondary Outcome: Acceptability as Measured by the tDCs Experience Questionnaire
Description: The tDCS experience questionnaire contains 10 questions based on a scale from 0-10, 0 being strongly disagree and 10 being strongly agree.
  Higher scores indicating greater acceptability for 7 questions and lower scores indicating greater acceptability for 3 questions resulting most desirable score of a 70.
Time Frame: week 3
Population: All participants completed tDCS experience questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 60 | 60
score on a scale | 62.93 (8.48) | 64.93 (9.66)

4. Secondary Outcome: Number of Participants With Possible Side Effects of Treatment
Description: If any side effects are reported, the degree of relatedness to the intervention will be assessed on a 10-point scale, from 0 (not at all) to 10 (to a high degree). The questionnaire ask to what extend did the participant experienced symptoms like, tingling, itching sensation, burning sensation, pain at the stimulation site, fatigue, nervousness, headache, difficulty concentrating, or mood change.
Time Frame: week 3
Population: Participants who experienced and reported any side effect.
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 60 | 60
Participants | 0 | 0

5. Secondary Outcome: Feasibility as Assessed by the Number of Participants That Complete the Full tDCS Protocol
Description: We will calculate the percentage of participants who a) meet the inclusion criteria, b) agree to be randomly assigned, c) complete the full tDCS protocol, and d) attend the follow-up assessment.
Time Frame: week 3
Population: All participants completed full tDCS protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 60 | 60
Participants | 60 | 60

ADVERSE EVENTS:
Time Frame: 3 weeks, from the first day of tDCS session to the last day.
Description: All participants are assessed for adverse events, but none observed.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 0/61 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04016272/Prot_SAP_001.pdf